CLINICAL TRIAL: NCT02702128
Title: Preventive EXACYL® on Perioperative Bleeding During Orthognathism of Maxillary Surgery
Acronym: LEFORTEXACYL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2014_68; 2015-002175-24 (EudraCT Number)
Record Dates: First submitted 2016-03-02; First posted 2016-03-08 (Estimated); Last update posted 2020-10-19 (Actual); Status verified 2020-03

CONDITIONS: Peri-operative Hemorrhage or Hematoma; Surgery; Retrognathism
Keywords: Bleeding perioperative; EXACYL; Oorthognathism surgery; Hematoma
MeSH Terms: conditions — Hematoma; Retrognathia | interventions — Tranexamic Acid; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tranexamic acid (Active Comparator): 1g of Tranexamic acid on 1hour and 1g of tranexamic acid on 8 hours
  Interventions: Drug: Tranexamic Acid
- saline solution (Placebo Comparator): 30mL of saline solution on 1 hour and 30mL of saline solution on 8 hours
  Interventions: Drug: saline solution

INTERVENTIONS:
Drug: Tranexamic Acid — 1g of tranexamic acid on 1 hour and 1g of tranexamic acid on 8 hours
  Arms: Tranexamic acid
Drug: saline solution — 30mL of saline solution on 1 hour and 30mL of saline solution on 8 hours
  Arms: saline solution

SUMMARY:
Prospective, randomized, double-blind, placebo-controlled, mono center, Phase III trial to compare EXACYL in preventive with placebo on perioperatory bleeding in orthognathism surgery.

DETAILED DESCRIPTION:
The aim of our study was to evaluate the clinical value of preventive treatment EXACYL® on bleeding during surgery to orthognathism. Our hypothesis is that this preventive treatment is not enough reduces bleeding to cause a change in patient management (count additional blood count, extra padding, transfusion).

Prospective equivalence trial type controlled by two parallel group, randomized, triple-blind (patient, surgical team, anesthesia team).

* EXACYL® Group: 1 syringe 1g EXACYL® on one hour + 1 syringe 1g EXACYL® on 8 hours
* Control group: 1 syringe 30 mL of saline on one hour + 1 syringe 30 mL saline on 8 hours Main criteria is amount of blood during the entire hospitalization: bleeding during surgery completed in the amount of blood present in the suction drains and nasogastric tube until ablation thereof.

ELIGIBILITY:
Inclusion Criteria:

* Patients to be operated on an osteotomy of the maxilla through a orthognathism surgery in the department of surgical specialties Salengro hospital
* Senior surgeon
* Hb ≥ 12 g / dL in the preoperative
* Patient ASA 1 or 2

Exclusion Criteria:

* Patient with coagulation disorders
* Patients treated with anticoagulant or antiplatelet
* Patients who require anticoagulation postoperatively
* Patient with against-indication to EXACYL® ( severe renal failure , convulsions history, history of thromboembolism venous or arterial )
* Surgery recognized preoperatively as particularly complicated by surgeons

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2016-01-03 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
bleeding perioperative | discharge from the hospital between 2 and 5 days
  bleeding during surgery and bleeding after surgery until hospitalization discharge

SECONDARY OUTCOMES:
bleeding during surgery | end of the surgery
  Amount of blood during surgery including : blood in the surgical aspiration, in compresses ( assessed by weighing compresses ) in the anesthetic aspiration (when extubation ) and the nasogastric tube at the end of surgery
EVA comfort surgery | end of the surgery
  Visual Analogue Scale for evaluation of surgical comfort
operative time | end of the surgery
  duration in minute of the surgery
Delta hemoglobin | Day 1 after surgery
  Difference between preoperative hemoglobin and postoperative ( Measured on the first preoperative and the second on the assessment conducted on Day 1)
EVA comfort patient | day 1 after surgery
  Visual Analogue Scale for assessment of patient comfort in day 1
Number of red blood cell transfused | discharge from the hospital between 2 and 5 days
  Number of red blood cell transfused
EVA fatigue patient | discharge from the hospital between 2 and 5 days
  visual analogue scale for assessment of the fatigue of the patient to the hospital discharge
Hospitalisation stay | discharge from the hospital between 2 and 5 days
  Hospitalization stay on day
Incidence of nausea and vomiting | discharge from the hospital between 2 and 5 days
  Incidence of nausea and vomiting calculated by the anti emetic dose received by the patient during hospitalisation
Thrombotic complications | discharge from the hospital between 2 and 5 days
  Number of thrombotic complications or cardiac complications during the hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Elsa Jozefowicz, MD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hôpital Roger Salengro, CHRU de Lille, Lille, France

IPD SHARING:
Plan to Share IPD: Undecided